CLINICAL TRIAL: NCT02123238
Title: Non-Supine Positioning in Treatment of Surgical Patients With Obstructive Sleep Apnea
Brief Title: Positioning of Surgical Patients With Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-14-549
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Other): standard of care positioning (0 degree)
  Interventions: Other: bed positioning
- 30 degree (Other): 30 degree bed positioning
  Interventions: Other: bed positioning
- 60 degree (Other): 60 degree bed positioning
  Interventions: Other: bed positioning

INTERVENTIONS:
Other: bed positioning

SUMMARY:
The study aims to evaluate the effect of non-supine positioning in the treatment of surgical patients with obstructive sleep apnea. The hypothesis is that non-supine positioning will result in a decrease in acute hypoxic events, defined as the number of apneas/hypopneas per hour of sleep.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial that will comprise of two stages. Stage 1 is a pilot study of 30 patients at high risk or diagnosed with obstructive sleep apnea who are scheduled for routine surgery. These patients will be randomized 1:1:1 to standard of care (0 degree bed angle), 30 degree bed angle, or 60 degree bed angle. Acute hypoxic events will be analyzed pre and post-op in the randomly assigned bed position. PACU nurses will also be surveyed for patient-favored non-supine positioning (30 vs. 60 degrees). Stage 2 will be a larger, powered trial to evaluate the efficacy of just one bed angle (30 or 60 degrees) based on the Stage 1 results.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 1 night postoperative hospital stay
* More than 18 and less than 80 years old
* Identified as high risk of OSA (SACS > 15) or a history of OSA without CPAP treatment

Exclusion Criteria:

* Unwilling or unable to give informed consent
* Undergoing nasal, eye, head/neck surgery, intracranial or cardiac/thoracic surgery
* Currently undergoing treatment for sleep apnea including CPAP
* Requiring prolonged postoperative ventilation
* NYHA functional class III and IV
* Valvular heart disease, dilated cardiomyopathy, implanted cardiac pacemaker, or unstable angina
* Myocardial infarction or cardiac surgery within 3 months
* Chronic obstructive pulmonary disease, or asthma
* Presence of tracheostomy, facial, neck, or chest wall abnormalities
* Abdominal aortic aneurysm surgery, chemotherapy, or immunosuppressive therapy within 3 months
* Visiting preoperative clinic less than 3 days before surgery
* Requiring postoperative nasogastric tube

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Acute Hypoxic Index (AHI) | 3 days
  study will look at the effect of bed positioning on Acute Hypoxic Index (AHI), which is defined as the number of apneas/hypopneas per hour of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Aryeh Shander, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States